CLINICAL TRIAL: NCT06345768
Title: Effect of Stress Ball Applied Before Cholecystectomy Surgery on Surgical Fear, Anxiety and Comfort of Patients: A Randomized Controlled Trial
Brief Title: The Effect of the Stress Ball Applied Before Colocystectomy Surgery on Patients; Surgical Fear, Anxiety and Comfort.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Scy123456789
Record Dates: First submitted 2024-03-23; First posted 2024-04-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cholecystitis; Stress; Fear; Comfort
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The researcher obtained 6 cm-diameter, moderate hardness, compressible balls made of silicone material in similar colors, mainly blue and green tones, some of which combined both colors featuring an Earth motif, before the study.
  Interventions: Other: Stress Ball
- Control group (No Intervention): Patients included in the control group had no intervention performed after completing the scale tools on the pretest, and 30 minutes later, the Surgical Fear Questionnaire, VAS-A and General Comfort Questionnaire were administered (posttest). Patients in the control group were not given stress balls for the pretest or posttest. No intervention was applied to patients in the control group. The scales were completed by researchers via face-to-face interviews in the preoperative waiting unit.

INTERVENTIONS:
Other: Stress Ball — The researcher obtained 6 cm-diameter, moderate hardness, compressible balls made of silicone material in similar colors, mainly blue and green tones, some of which combined both colors featuring an Earth motif, before the study. After patients in the intervention group applied the scale tools in the pretest, the intervention stage began. Patients were given stress balls. When patients were given information about the stress ball application, they were called squeeze balls with the aim of not inferring that the process was stressful. The participants were given the right to choose the stress ball (color and pattern preference). Patients were taught to count from one to three and to squeeze and relax the ball and were told to continue in this way until the end of the intervention. Additionally, they were requested to pay attention to the squeeze ball and squeeze with focus. The participants were asked to repeat this process for a total of 30 minutes, and the researcher remotely observed
  Arms: Intervention

SUMMARY:
Cholecystectomy is the most common major abdominal surgical procedure in western countries. Patients may experience fear and anxiety before surgery.

Stress ball, one of the distraction methods, is an effective method in providing cognitive focus. It is seen that the stress ball method is used to reduce patients' anxiety and pain. Squeezing the stress ball during the surgical procedure allows patients to have direct control over the object, increasing their sense of empowerment. In this way, it has a positive effect on anxiety and patient satisfaction without interfering with the surgical procedure.

In this study, it is aimed to evaluate the effect of preoperative use of stress ball on patients' fear, stress and comfort in order to determine the effect of stress ball applied before cholecystectomy surgery on patients' surgical fear, stress and comfort. It is thought that the data obtained as a result of the research will provide evidence for the effect of the stress ball, which is a non-pharmacological method used before the procedure, on fear, stress and comfort.

DETAILED DESCRIPTION:
This study was planned to examine the effect of a stress ball applied to patients before laparoscopic cholecystectomy on preoperative anxiety, surgical fear and comfort. Patients were given a stress ball before the procedure, and the other group received routine care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to speak and understand Turkish
3. Being literate
4. Patients who underwent elective laparoscopic cholecystectomy
5. Volunteering to participate in the study

Exclusion Criteria:

1. Use of any analgesic or anxiolytic preoperatively
2. Any physical obstacle to using a stress ball (patients with partial paralysis or weak hand muscles)
3. History of psychiatric disorders or ongoing psychiatric treatment.
4. Emergency surgery
5. Open cholecystectomy
6. Hearing or perception problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Fear of surgery | 30 minutes before surgery
  The scale consists of 8 items and is an 11-point Likert type, with each item scored between 0 (I am not afraid at all) and 10 (I am very afraid). bottom of scale The lowest score that can be obtained from the dimensions is 0, the highest score is 40, the lowest score that can be obtained from the total scale is 0 and the highest score is 80.
Fear of surgery | Just before surgery
  The scale consists of 8 items and is an 11-point Likert type, with each item scored
Comfort | 30 minutes before surgery
  The scale contains a total of 48 items in four/six point Likert type; Four-point Likert type was preferred due to its ease of use. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48.
Comfort | Just before surgery
  The scale contains a total of 48 items in four/six point Likert type; Four-point Likert type was preferred due to its ease of use. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48.
Stress | 30 minutes before surgery
  It was designed by researchers similar to the use of "Visual Analog Scale (VAS)". VAS is used to make measurable some values that cannot be measured numerically, which are evaluated by individuals by marking on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end indicates that the individual is "very bad".
Stress | Just before surgery
  It was designed by researchers similar to the use of "Visual Analog Scale (VAS)". VAS is used to make measurable some values that cannot be measured numerically, which are evaluated by individuals by marking on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end indicates that the individual is "very bad".

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Merve Alptekin, Principal Investigator — Kocaeli University
Locations (1):
- Samsun Üniversitesi Klinik Araştırma Etik Kurulu, Samsun, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No